CLINICAL TRIAL: NCT03125161
Title: A Prospective, Randomized, One-center Study Comparing Hepatic Arterial Infusion Plus Chemotherapy ± Target Therapy and Chemotherapy ± Target Therapy Alone in Patients With Unresectable Colorectal Cancer Liver Metastases
Brief Title: Study Comparing HAI Plus Chemotherapy and Chemotherapy Alone in Patients With Unresectable CRLM
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Prof., Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HAICRLM
Record Dates: First submitted 2017-04-19; First posted 2017-04-24 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Colorectal Adenocarcinoma Metastatic to the Liver
Keywords: colorectal cancer; liver metastasis; hepatic arterial infusion; chemotherapy; target therapy; conversional resection rates
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): HAI plus chemotherapy ± target therapy
  Interventions: Drug: HAI; Drug: chemotherapy ± target therapy
- Arm B (Active Comparator): chemotherapy ± target therapy
  Interventions: Drug: chemotherapy ± target therapy

INTERVENTIONS:
Drug: HAI — HAI
  Arms: Arm A
Drug: chemotherapy ± target therapy — chemotherapy ± target therapy

SUMMARY:
To date no prospective trials have been completed that demonstrated whether HAI is an effective adjunct to systemic chemotherapy (target therapy) with respect to advantages in conversional resection rates and survival compared with chemotherapy (target therapy) alone. The primary objective of this trial is to determine conversional resection rates and survival for patients with colorectal cancer liver metastasis are treated with HAI plus chemotherapy ± target therapy, compared to chemotherapy ± target therapy only.

ELIGIBILITY:
Inclusion Criteria:

* All patients must meet the following criteria:
* Patients must have histologically confirmed incurable CRLM and no clinical or radiographic evidence of extrahepatic disease
* Patients is medically eligible to receive HAI, as determined by the MDT (multidisciplinary team)
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
* Age > 18 years
* Subject life expectancy > 3 months
* Platelets > 100×103/mm3
* Total bilirubin <1.5mg/dl
* Creatinine level < 2.0 mg/dl
* All patients must sign an informed consent form

Exclusion Criteria:

* The CRLM is amenable to curative surgical therapy
* Prior radiation, TACE or HAI to the liver
* Uncorrectable coagulopathy
* Subject is pregnant, nursing, or wishes to become pregnant during the study Other serious medical condition (uncontrolled infection, uncontrolled cardiac disease) would preclude study treatment or impact survival
* Current or planned treatment with any experimental chemotherapy or target drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-04-30 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
conversional resection rates | 2-4 months

SECONDARY OUTCOMES:
overall response rates | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Xu, PhD, Study Chair — Fudan University
Locations (1):
- Zhongshan hosptial, Fudan University, Shanghai, China